CLINICAL TRIAL: NCT01447758
Title: Safety, Tolerability and Pharmacokinetics of LEO 29102 Cream in Atopic Dermatitis. A Multicentre, Prospective, Randomised Phase Ib Study in Subjects Investigating Safety,Tolerability and Pharmacokinetics of LEO 29102 Cream (2.5 mg/g) When Treating Atopic Dermatitis Lesions Twice Daily for 7 Days (Cohorts I, II and III) and 6 Weeks (Cohort IV)
Brief Title: Safety, Tolerability and Pharmacokinetics of LEO 29102 Cream in Atopic Dermatitis.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LEO 29102-C26
Record Dates: First submitted 2011-07-13; First posted 2011-10-06 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2013-04

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — 2-(6-(2-(3,5-dichloro-4-pyridyl)acetyl)-2,3-dimethoxyphenoxy)-N-propylacetamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LEO 29102 2,5 mg/g cream (Experimental)
  Interventions: Drug: LEO 29102
- LEO 29102 Cream Vehicle (Placebo Comparator)
  Interventions: Drug: LEO 29102 Cream Vehicle

INTERVENTIONS:
Drug: LEO 29102 — Cream, 1,7mg/cm2 BSA, BID, 7 days In Cohort I, II and III, 6 weeks in Cohort IV
  Arms: LEO 29102 2,5 mg/g cream
Drug: LEO 29102 Cream Vehicle — Cream, 1,7mg/cm2 BSA, BID, 7 days in Cohort I and II, 6 weeks in Cohort IV
  Arms: LEO 29102 Cream Vehicle

SUMMARY:
The purpose of this Phase Ib study is to investigate the safety, tolerability and pharmacokinetics of LEO 29102 2,5 mg/g cream when treating atopic dermatitis (AD) lesions from 10 up to 100% of the body surface area (BSA) twice daily (BID) for 7 days (Cohorts I, II, III) and from 10% up to 50% of BSA (bid) for 6 weeks (Cohort IV). This trial will be performed in four cohorts. Cohort I, II and III includes patients with a larger BSA that increases from one cohort to the next. After each cohort (Cohort I, II)a blinded evaluation of the safety and tolerability data will assess whether a stepwise increase in the percentage of "to be treated BSA" is justified. Cohort IV will start dosing after finalisation of Cohort II and after submission of data from Cohort I and II to the national authority and IEC for review.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of AD defined according to Hanifin and Rajka.
2. Investigator Global Assessment scored as mild (2) to severe (4) AD.
3. At screening, AD lesions amenable for treatment involving 10% to < 25% (Cohort I), 25% to < 50% (Cohort II), 50% to 100% (Cohort III) and 10% to < 50% (Cohort IV) of the total BSA.
4. On Day -1, AD lesions amenable for treatment involving 10% to < 28% (Cohort I), 25% to < 55% (Cohort II), 50% to 100% (Cohort III) and 10% to < 55% (Cohort IV) of the total BSA.
5. Adult male or female subjects, aged 18 to 65 years, inclusive.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2011-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
PK profile - Cohort I, II, III | Predose, 1h, 2h, 4h, 6h, 12h, 13h, 14h, 16h, 18h, 24h (on day 1 and 7) and 36h, 48h, 72h (on day 7 only)
  Cmax, AUC, Tmax
Tolerability and safety of LEO 29102 cream - Cohort I, II, III | 14 Days
  Number of subjects with AEs and change from baseline in vital signs (blood pressure, pulse rate, respiratory rate body temperature), ECG parameters, clinical laboratory, physical examination
PK profile - Cohort IV | Day 1, 14, 28, 42: Pre AM dose and 1h, 2h, 4h, 6h, 12h. Post AM dose, but prior to PM dose and 24 h, 36h, 48h, 72h after AM dose Day 42
  Cmax, AUC, Tmax
Tolerability and safety of LEO 29102 cream - Cohort IV | 49 Days
  Number of subjects with AEs and change from baseline in vital signs (blood pressure, pulse rate, respiratory rate body temperature), ECG parameters, clinical laboratory, physical examination, SCORAD, EASI and IGA by stratum, treatment and visit.

SECONDARY OUTCOMES:
Dermis concentration of LEO 29102 and its metabolites LEO 28386 and LEO 26989 after multiple topical applications in subjects with AD (Cohorts II and IV, Subgroup 1) | 10 Days for cohort II; 42 days for cohort IV, subgroup 1
Biomarkers in AD lesions before and after multiple topical applications in subjects with AD (Cohorts I and IV, Subgroup 2) | 10 Days for cohort I, 42 days for cohort IV, subgroup 2

CONTACTS AND LOCATIONS:
Overall Officials: Diamant Thaci, MD, Principal Investigator — Goethe University
Locations (8):
- Germany (8):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Klinik und Poliklinik für Dermatologie und Allergologie der Universität Bonn, Bonn
  - Universitätshautklinik Essen, Essen
  - Department of Dermatology, Johann Wolfgang Goethe-University, Frankfurt am Main
  - SRH Wald-Klinikum Gera gGmbH, Gera
  - Clinical Trial Center North, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitätshautklinik Münster, Münster

IPD SHARING:
Plan to Share IPD: No